CLINICAL TRIAL: NCT05223608
Title: Prospective Cohort With Clinic-biologic Database of Patients Treated by Immunotherapy
Acronym: ImmuCCo
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Oscar Lambret (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ImmuCCo-1905
Record Dates: First submitted 2022-01-24; First posted 2022-02-04 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Solid Tumor, Adult
Keywords: Prospective cohort; Clinic-biologic database; Solid tumor; Immunotherapy

STUDY DESIGN:
Intervention Model Description: Observational study model with additional blood samples and urine collection
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- ImmuCCo Cohort (Other): Blood sampling at initiation of immunotherapy, at the first tumor assessment, in case of severe toxicity.
  Urine collection at initiation of immunotherapy.
  Interventions: Other: ImmuCCo Cohort

INTERVENTIONS:
Other: ImmuCCo Cohort — Blood sampling at initiation of immunotherapy, at the first tumor assessment, in case of severe toxicity. Urine collection at initiation of immunotherapy.

SUMMARY:
ImmuCCo-1905 is a monocentric interventional study on patients treated by immunotherapy, which consist in establishment of a prospective clinic-biologic database over 5 years, associated with a biobank. This database will allow carrying out works aiming at assessing immunotherapy in real life situation.

DETAILED DESCRIPTION:
The aim of this study is to establish a prospective clinic-biologic database of patients treated by immunotherapy. This database will allowed to carry out works (such as translational research) aiming at assessing immunotherapy in real life situation.

Other objectives of the study include:

* Describe overall survival, progression-free survival, response to immunotherapy (in particular hyper-progression, pseudo-progression) considering the first tumor assessment and the best response, prolonged response
* Identifying prognostic factors of overall survival, progression-free survival, hyper-progression, best response under immunotherapy
* Describe AEs (Adverse Events) potentially associated with immunotherapy, their kinetics of appearance, from the start of treatment and after the end of treatment in order to assess the risk of delayed appearance
* To identify factors associated with increased risk of severe adverse event (grade > 2 or leading to end of treatment) potentially related to immunotherapy, from the beginning of immunotherapy to 1 year after this start of the treatment, in patients who received at least 4 doses or who stopped the treatment earlier (before 4 doses) due to toxicity.
* Identifying delayed adverse events potentially related to immunotherapy, occurring between 90 days and 1 year after the treatment discontinuation, in patients who received at least 4 doses or who stopped the treatment earlier (before 4 doses) due to toxicity.
* To identify and describe rare toxicities
* To evaluate the association between co-medications and disease evolution
* To evaluate the association between co-medications and toxicities occurrence

Translational research objectives:

* To identify biomarkers that might be associated with tumor response and/or toxicity of immunotherapy from:

  * Establishment of serum and plasma bank which will be used for diverse works;
  * A systematic analysis of the lymphocyte profile
* To study the impact of tabagism on efficacy and toxicity of immunotherapy from systematic collection of urinary cotinine.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Beginning a first immunotherapy by immune checkpoint inhibitor - anti-PD1 (Programmed cell Death protein-1), anti-PDL1 (Programmed cell Death protein-1 ligand), anti-CTLA4 (Cytotoxic T-Lymphocyte associated protein 4), as monotherapy or in combination, in the Centre Oscar Lambret (COL)
* In neo-adjuvant, adjuvant, recurrence or metastatic situation
* Suffering from solid tumor histologically documented
* Signed written informed consent
* Patient covered by the French " "Social Security" regime If the patient is already enrolled in clinical trial involving immunotherapy, the agreement of the sponsor of this new trial will be sought before his/her inclusion.

Exclusion Criteria:

* Pregnant or breastfeeding women
* Patient already treated by immunotherapy by immune checkpoint inhibitor
* Person under guardianship
* Inability to comply with medical follow-up of the trial (geographical, social or psychic reasons)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2022-03-03 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Number of patients treated by immunotherapy and registered in the database. | 5 years
  Number of patients treated by immunotherapy and registered in the database

SECONDARY OUTCOMES:
Overall Survival | 6 years
  Time between date of start of immunotherapy to date of death whatever the cause. Patients alive at last follow-up will be censored.
Progression-Free Survival | 6 years
  Time between start of immunotherapy to date of disease progression or death whatever the cause. Alive, non-progressive patients at last follow-up will be censored.
Tumor response | 6 years
  Tumor response will be based on the first tumor assessment performed during the immunotherapy. Objective response according to iRECIST (Response Evaluation Criteria in Solid Tumours for immunotherapy) criteria will be defined at the first tumor assessment and during the course of the treatment, meaning until disease progression of start of another systemic treatment.
  Responses will be: Complete response (iCR), partial response (iPR), stability (iSD), progression, or pseudo-progression. Confirmed progressive disease (iCPD) will be distinguished from pseudo-progression (iUPD) according to control images. Hyper-progression will be defined as a progression according to iRECIST criteria and a doubling of tumor growth rate.
  A prolonged tumor response will be defined as a progression free survival duration at least 3 time superior to median duration of progression free survival of patients of the study presenting the same disease.
Co-medications | 6 years
  All comedications given during the course of the study will be compiled
Toxicity of immunotherapy | 6 years
  All Adverse events occuring from the start of the immunotherapy to the follow-up performed on year after the end of the immunotherapy will be notified, whatever the grade and the relationship with immunotherapy, apart from those undoubtfully related to the disease or the progression of the disease.The AE will also be notified in case of start of a second line of treatment, apart from thos undoubtfully related to this second line of treatment. The main analysis will be done on AE potentially related to immunotherapy. The relationship will be evaluated by a medical expert of immunotherapy. AE will be graded according to CTCAE v5.0 classification. Patients who received less than 4 doses will be considered non-evaluable for this outcome apart from those who discontinued treatment because they had a toxicity. Each AE with a grade > 2 and/or leading to treatment discontinuation will be considered as severe.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra FORESTIER, MD, Principal Investigator — Centre Oscar Lambret
Locations (1):
- Centre Oscar Lambret, Lille, Hauts-de-France, France

IPD SHARING:
Plan to Share IPD: No